CLINICAL TRIAL: NCT02261311
Title: An Innovation During the Surgical Wait; Evaluation of the Opportunity for Intervention
Acronym: RADSII
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20130232-01H
Record Dates: First submitted 2014-09-25; First posted 2014-10-10 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
Keywords: Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Additional tissue samples will be collected at the time of initial biopsy. The samples will be stored for neoadjuvant studies that the patient may choose to participate in during the wait time between diaganosis and surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quality of Life, tissue collection: All participants will complete the GAD-7 and Cancer Locus of Control Scale - Course of Illness Subscale questionnaires and additional tissue will be collected at the time of the diagnostic biopsy.
  Interventions: Other: Quality of Life

INTERVENTIONS:
Other: Quality of Life — All participants recruited will complete a questionnaire prior to their breast biopsy and then again approximately one week before their surgery. The questionnaire is focused on the level of anxiety patients experience during the wait time between diagnosis and surgery. Additional tissue will be collected at the time of the diagnostic biopsy.

SUMMARY:
The investigators will compare the differences in the scores between the baseline questionnaire (at diagnosis) and the second questionnaire (at treatment) in the RADS II patients that enrolled in pre-treatment trials versus those that don't.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Diagnosis of BI-RADS 4 and 5 (highly suspicious for carcinoma) on an initial imaging
* >2cm area of disease
* Provide informed consent

Exclusion Criteria:

* Previous neo-adjuvant therapy
* Patients with recurrent disease

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with BIRADS 4/5 on initial mammogram.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-03; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life | up to 6 weeks
  To determine if there are improvements in the measurements of anxiety through quality of life questionnaires completed at 2 different time points when participating in a window of opportunity trial verses not participating in a window of opportunity trial.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arnaout, Surgeon, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada